CLINICAL TRIAL: NCT06475287
Title: The Efficacy and Safety of HAIC Combined With TQB2450 and Anlotinib in Second-line Treatment of Advanced Hepatocellular Carcinoma: an Open, Single Arm Exploratory Study
Brief Title: HAIC Combined With TQB2450 and Anlotinib in Second-line Treatment of Advanced Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Chief physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2403292-20-2405A
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC combined with TQB2450 and Anlotinib (Experimental)
  Interventions: Drug: HAIC（Mitoxantrone+Raltitrexed）、anlotinib、TQB2450

INTERVENTIONS:
Drug: HAIC（Mitoxantrone+Raltitrexed）、anlotinib、TQB2450 — The combination therapy of HAIC with TQB2450 and Anlotinib was administered to enrolled patients in no particular order. Patients received routine hepatic artery catheterization via femoral artery puncture, followed by routine hepatic artery catheterization and infusion chemotherapy with 5% sodium bicarbonate 150ml + liposomal mitoxantrone (10mg) for 2-4 hours + Raltitrexed (2mg/m2) for 2-4 hours, every three weeks for at least two cycles. Systemic treatment was given every 21 days, with a fixed dose of 1200mg of TQB2450 injection on the first day of each systemic treatment cycle (1-7 days after HAIC treatment), administered intravenously over 60 minutes initially, followed by 30 minutes if tolerated. Anlotinib was administered orally once daily at a dose of 10mg, with a two-week break every three weeks. Treatment continued until unacceptable toxicity or loss of clinical benefit (as assessed by the investigator based on imaging, biochemical indicators, and patient clinical status).

SUMMARY:
Overall, although there are many options for second-line treatment of liver cancer, the ORR is mostly limited to within 20-30%, with a median PFS of 3-5 months and a median OS of 10-20 months. The overall situation is still unsatisfactory, with low objective tumor response rates and targeted immune resistance being the main reasons affecting treatment efficacy. Increasing local treatment or overcoming resistance is currently a hot research topic. The aim of this study is to explore the effectiveness and safety of HAIC combined with TQB2450 and anlotinib for second-line treatment of advanced HCC patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female aged 18-80 years or older;
* Diagnosed as advanced hepatocellular carcinoma (HCC) by histology, cytology, or clinical examination;
* Signed informed consent form
* The patient has received first-line treatment for hepatocellular carcinoma and the treatment has failed or is intolerable;
* Previously received HAIC treatment containing platinum;
* Early treatment allows for receiving tyrosine kinase inhibitor (TKI) treatment or bevacizumab treatment;
* Allow to receive immunotherapy in the early stage;
* At least one measurable lesion (according to RECIST 1.1 standard);
* Tumor tissue samples before treatment (if available)；
* Child Pugh A grade or ≤ 7 B grade within 14 days prior to enrollment;
* HIV antibody test result was negative during screening
* HIV antibody test result was negative during screening
* Any acute, clinically significant treatment-related toxicity (caused by previous treatment) must have been alleviated to ≤ 1 level before enrollment in the study, except for hair loss
* Patients with active hepatitis B virus (HBV) infection: HBV DNA<2000IU/mL obtained within 28 days before starting the study treatment, and received at least 7 days of anti HBV treatment (according to local standard treatment, such as entecavir) before joining the study, and were willing to continue to receive treatment during the study period; Patients with active hepatitis C virus (HCV) infection: HCVRNA<2000IU/mL obtained within 28 days prior to the start of study treatment, and who have received at least 7 days of anti HCV treatment before enrollment in the study and are willing to continue treatment during the study period

Exclusion Criteria:

* Previously received treatment with mitoxantrone;
* History of soft meningitis;
* Current or past autoimmune diseases or immunodeficiencies;
* Idiopathic pulmonary fibrosis, organizing pneumonia (such as bronchiolitis obliterans), drug-induced pneumonia or idiopathic pneumonia, or evidence of active pneumonia can be seen on screening chest computed tomography (CT) images. Allow radiation zone (fibrosis) to have radiation induced pneumonia;
* Known active tuberculosis;
* Within 3 months prior to the start of the study treatment, there was a significant cardiovascular disease, unstable arrhythmia, or unstable angina;
* History of congenital long QT syndrome or corrected QT interval during screening>500ms ;
* History of electrolyte disorders such as uncorrectable serum potassium, calcium, or magnesium;
* Received major surgical treatment within 4 weeks prior to the start of the study (excluding diagnosis) or expected to undergo major surgical treatment during the study period;
* Previously diagnosed with malignant tumors other than HCC within the 5 years prior to screening, excluding those with negligible risk of metastasis or death (e.g. 5-year OS rate>90%), such as fully treated in situ cervical cancer, non melanoma skin cancer, localized prostate cancer, in situ or stage I uterine cancer;
* Within 4 weeks prior to the start of the study treatment, there was a severe infection, including but not limited to hospitalization due to complications such as infection, bacteremia, or severe pneumonia;
* Administer therapeutic antibiotics orally or intravenously within 2 weeks prior to starting the study treatment. Patients who receive prophylactic antibiotics (such as preventing urinary tract infections or exacerbation of chronic obstructive pulmonary disease) are eligible to participate in the study;
* Previous allogeneic stem cell or solid organ transplantation;
* Received attenuated live vaccine treatment within 4 weeks prior to the start of the study, or expected to receive such vaccine during PD-1 monoclonal antibody treatment or within 5 months after the last dose of PD-1 monoclonal antibody;
* Untreated or incompletely treated esophageal and/or gastric varicose patients with accompanying bleeding or high risk of bleeding;
* Simultaneously infected with HBV and HCV;
* Symptomatic, untreated, or gradually progressing central nervous system (CNS) metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 24 months
  The proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time, including complete response and partial response

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China